CLINICAL TRIAL: NCT07160907
Title: The Impact of Elderly Simulation Experience on Aging Knowledge, Attitudes, Empathy, Communication Skills and Learning Satisfaction for Facility Care- Workers in Long-term Care Institutions : An Action Research and Effectiveness Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Jo Han Chung, researcher, Tzu Chi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: YLH-IRB-11418
Record Dates: First submitted 2025-06-26; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Careworker; Education
Keywords: Ageing Knowledge; Attitude; Empathy; Communication Skills; Learning Satisfaction
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: cluster randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this group will receive a comprehensive ageing simulation training program, which includes: (1) an ageing knowledge and empathy-focused lecture incorporating interactive videos and scenario-based video discussions; (2) an ageing simulation activity using the "PengZu Suit" to mimic physical decline across five caregiving scenarios; and (3) a peer group discussion facilitated by empathy-trained professionals. This intervention aims to enhance participants' ageing knowledge, care attitudes, empathy, communication skills, and learning satisfaction.
  Interventions: Behavioral: Ageing Simulation Experience Program
- Control group (Active Comparator): Participants in this group will receive only the ageing knowledge lecture, which includes basic concepts of aging and empathy delivered through multimedia materials. They will not participate in the simulation activity or the peer discussion session.
  Interventions: Behavioral: Ageing Simulation Experience Program

INTERVENTIONS:
Behavioral: Ageing Simulation Experience Program — Ageing Simulation Experience Program is a structured training that includes a multimedia lecture, a hands-on aging simulation using the PengZu Suit, and a peer discussion. It aims to enhance care workers' aging knowledge, empathy, attitudes, and communication skills through experiential learning.

SUMMARY:
This study aims to evaluate the effectiveness of an aging simulation experience course in enhancing the aging knowledge, care attitudes, empathy, communication skills, and learning satisfaction of care service personnel working in residential long-term care institutions.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effectiveness of an aging simulation experience course in improving aging knowledge, care attitudes, empathy, communication skills, and learning satisfaction among care workers in long-term care institutions. A total of 162 participants will be randomly assigned to an experimental group receiving an aging knowledge lecture, a hands-on aging simulation using aging suits, and a peer discussion session, or to a control group receiving only the lecture. Outcomes will be assessed before the intervention, and one and two months after. Both quantitative and qualitative analyses will be conducted to measure training effectiveness and inform future caregiver education programs.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be care workers currently employed at residential long-term care institutions in Eastern Taiwan, aged between 20 and 70 years. They must have at least one month of work experience in their current role, be literate, capable of completing written questionnaires, able to communicate in Mandarin or Taiwanese, and willing to provide informed consent to participate in the study.

Exclusion Criteria:

* Individuals will be excluded if they do not meet the above inclusion criteria, decline to participate or withdraw consent during the study, or are physically unable to safely engage in the aging simulation activity due to health or mobility limitations.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Aging Knowledge | baseline, month 1、2
  knowledge about Aging
Attitudes | baseline, month 1、2
  attitudes towards aging
Empathy | baseline, month 1、2
  Empathy for Aging
Communication Skills | baseline, month 1、2
  Communication Skills for Aging
Learning Satisfaction | baseline, month 1、2
  Learning satisfaction after class

CONTACTS AND LOCATIONS:
Locations (1):
- Tzu Chi University, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No